CLINICAL TRIAL: NCT05257681
Title: Inter-lobar Fissure Completion as a Salvage Treatment in Patients With Failed Bronchoscopic Lung Volume Reduction
Brief Title: Inter-lobar Fissure Completion in Patients With Failed Bronchoscopic Lung Volume Reduction
Acronym: SAVED-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Adnan Majid, MD, Chief Interventional Pulmonology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000048
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Emphysema or COPD
Keywords: COPD; Chronic Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease; Emphysema; Video-assisted thoracic surgery
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This study is expected to enroll a total of 20 subjects with a follow-up period of 3 months. All interventions and follow-up will be performed at the BIDMC. In current medical practice, emphysema patients that fail to achieve target lung volume reduction after endobronchial valves placement, are continued on current medical management for their COPD, with consideration for lung transplantation should they be eligible depending on clinical circumstances and degree of lung function impairment. The investigators plan to offer this patient population the possibility to undergo a VATS fissure completion and adhesiolysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fissure completion and adhesiolysis arm (Experimental): Patients will undergo a VATS or robotic interlobar lung fissure completion with pleural adhesiolysis. After a 3 month follow-up period, patients will fill additional quality of life questionnaires including the St.George Respiratory Questionnaire, COPD Assessment tool, and the modified medical research council dyspnea scale. Pulmonary function testing and a high-resolution CT scan will be performed at the end of the 3-month postoperative follow-up.
  Interventions: Procedure: Interlobar fissure completion and pleural adhesiolysis

INTERVENTIONS:
Procedure: Interlobar fissure completion and pleural adhesiolysis — A video-assisted thoracic surgery or robotic approach will be used to perform pleural adhesiolysis and the lobar fissure adjacent to the previously targeted lobe during bronchoscopic lung volume reduction will be completed using a surgical stapler.

SUMMARY:
The purpose of this protocol is to perform a pilot prospective controlled clinical trial to evaluate the potential role of lung fissure completion with pleural adhesiolysis strategy (experimental intervention) in severe emphysema/COPD patients with failed bronchoscopic lung volume reduction (BLVR) via the use of endobronchial valves (EBVs) therapy. In select patients, the lung fissure completion with adhesiolysis strategy will be performed by video-assisted thoracoscopic surgery (VATS) guided stapling along the lung fissures to reduce collateral ventilation with adhesions removal and determine whether this experimental strategy will improve outcomes after failed BLVR in patients with severe emphysema/COPD.

DETAILED DESCRIPTION:
The investigators will approach all patients with failed EBV therapy. Patients with less than 350 ml of volume reduction in the target lobe and persistent dyspnea [score greater or equal to 2 on the Modified Medical Research Council Dyspnea Scale (mMRC)] after EBV placement will be considered to have failed EBV therapy due to adhesions or collateral ventilation being present. Only patients with failed EBV therapy will be approached to participate in our study. Once the patient agrees to participate and sign the consent, all the screening information collected as part of the standard of care will be extracted retrospectively from the medical records including appointment details, 6MWD, and PFTs results. In addition, during the same visit, health-related quality of life will be measured using the Saint George Respiratory Questionnaire (SGRQ) and COPD Assessment Test (CAT), and dyspnea will be assessed with the self-reported mMRC.

VATS Inter-Lobar Fissure Completion and Pleural Adhesiolysis The clinician providing general anesthesia will be familiar with thoracic anesthesia and complications in patients with severe COPD undergoing thoracic surgery and endoscopic valve implantation. Total IV anesthesia will be used during all bronchoscopic procedures. Routine antimicrobial prophylaxis will be administered at induction. The antimicrobial choice will be based on the subject's allergies and/or history of resistant organisms.

The experimental procedure will be performed via VATS under inhaled anesthetic agents by an experienced thoracic surgeon from BIDMC. The clinician providing general anesthesia will be familiar with thoracic anesthesia and complications in patients with severe COPD undergoing thoracic surgery and endoscopic valve implantation. A double-lumen endotracheal tube will be inserted allowing one-lung ventilation and the maximal collapse of the operative lung. The subject will be placed in lateral decubitus with the operative side up. Disinfection of the surgical site will be performed with the application of an antiseptic solution and the subject will be draped in the usual sterile fashion. The thoracic surgeon will perform multiple rib blocks and inject the skin incisions with bupivacaine. Through small incisions, the surgeon will create a camera port through the intercostal space and then the anterior and posterior inferior ports. Electrocautery will be used for adhesion release of the ipsilateral lung of the target lobe. Dissection and exposure of the anterior aspect of the hilum will then be performed using electrocautery. Following the exposure, stapling will be performed on the incomplete fissure adjacent to the target lobe, using the Endo GIATM (CovidienTM, Mansfield, MA) FDA-approved surgical stapler. The lung tissue will be dissected until the pulmonary artery is seen, in a similar fashion to the method used in lobectomies and segmentectomies. Multiple surgical stapler activations will be used to complete the target fissure along the fissure line.

An attempt at conversion to a complete fissure will be made, though depending on the anatomy, it may be possible that residual incomplete fissure of up to 5% may be tolerated. Hemostasis will be evaluated. Sterile water will then be used to fill the surgical area, followed by lung inflation and inspection to verify for air leaks at the level of the stapling. If an air leak is detected, suturing, re-stapling, or applying pleural sealants will be used to seal it. The patient will be monitored closely for air leaks in the postoperative setting in case there is the persistence of the air leak despite the measures taken and valve presence, a second intervention will be considered based on the thoracic surgeon's judgment. Once the fissure is surgically completed, a chest tube will be placed and connected to a chest drainage system.

In the setting that the thoracic surgeon will not be able to complete the fissure up to 95% due to anatomic restraints, the procedure will then be ended without valve implantation, as the presence of residual collateral ventilation is expected. All patients will receive standard of care post-operative management, and subjects will continue to be followed for any procedure-related adverse events until the event has subsided or, in case of permanent impairment, until the event stabilizes, and the overall clinical outcome has been ascertained. At that time, the subject will be withdrawn from the study and will be considered as an "Enrollment Failure" and recorded as such for statistical analysis.

Bronchoscopic Evaluation The double-lumen endotracheal tube will be removed, and a single-lumen tube (8.0 to 8.5 mm) inserted. The lung will be completely re-inflated before this evaluation to return them to normal anatomy.

Flexible bronchoscopy will be done by the interventional pulmonologist. The bronchoscope will be passed via the endotracheal tube and the major airways will be examined. The placement of the EBVs will be assessed. In case one of the valves is not adequately placed, the interventional pulmonologist will adjust it. If any valve needs to be replaced, the replacement will be performed at this point. A bronchial wash will be performed with samples sent for culture. If there are unexpected findings, such as a lesion suspicious for carcinoma or secretions suggesting infection, then appropriate clinical samples will be obtained, and the subject will be re-evaluated, the study team will then determine if the subject will be withdrawn from the study and will be considered as an "Enrollment Failure" and recorded as such for statistical analysis.

Postoperative Persistent Air-Leak Management In the setting of a persisting air-leak > 5 days after the procedure, the investigator will proceed to the removal of the most proximal valve from the treated lobe (if the left upper lobe is the treatment lobe, the removal will be from a lingular segment). If there is a resolution of the air leak within 48 hours, replacement of the valve will be considered and scheduled in 6 weeks. During the valve replacement procedure, if previously placed valves are observed to be sub-optimally placed, the investigator may remove and replace any sub-optimally placed valves.

If the air leak does not resolve within 48 hours after the first valve removal, all remaining valves will be removed. In the setting of a persistent air-leak despite previous interventions, further management will be based on the investigator's judgment and per standard of care (chemical pleurodesis or conservative management). Chest tube maintenance > 7 days in presence of a persistent air leak will also be considered as a thoracic serious adverse event and recorded in the AE CRF as part of the study's safety evaluation.

The management algorithm for persistent air-leaks was adapted from the expert consensus by Valipour et al. Clinical management of persistent air-leaks may vary depending on clinical circumstances, so exceptions to these guidelines will not be considered protocol deviations.

Pneumothorax Management Pneumothorax after valve placement can be an effect of the desired treatment response that is associated with complete lobe treatment and atelectasis. The management of pneumothorax is an integral part of the treatment. The origin is thought to be from the rupture of stretched diseased tissue that is adjacent to the volume reduced lobe. Management for pneumothorax associated with EBVs will be conducted according to expert consensus and our internal algorithm, which represents standard-of-care for pneumothorax management.

Follow-up Period After VATS fissure completion and adhesiolysis, patients will be placed on a standardized follow-up protocol used for individuals that underwent video-assisted thoracic surgery. Data from follow-up appointments at 14 days and 3 months will be collected from the medical records retrospectively including appointment details, complications, CT-scan results, 6MWD, and PFTs results. Target lung volume reduction (TLVR) will be assessed at 3 months using the CT scans performed on patients as part of their standard of care. The only procedures that will be considered research after the initial surgical intervention would be the measurement of health-related quality of life with the SGRQ and CAT, and dyspnea assessment with the self-reported mMRC at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years.
* Stable with less than 10mg prednisone (or equivalent) daily.
* Nonsmoking for 4 months prior to screening and willing to not smoke during the study duration.
* Current pneumococcus vaccination.
* Current influenza vaccination.
* Target lung volume reduction <350ml after bronchoscopic lung volume reduction (BLVR).
* Persistent dyspnea defined as an mMRC score greater or equal to 2 after bronchoscopic lung volume reduction (BLVR).
* Endobronchial valves (EBV) are still in place.
* Willing and able to complete protocol required study follow-up assessments and procedures.

Exclusion Criteria:

* Clinically significant (greater than 4 tablespoons per day) mucus production.
* Myocardial infarction within 6 months of screening.
* Decompensated heart failure.
* Three or more pneumonia episodes in last year.
* Three or more COPD exacerbation episodes in the last year.
* Prior lung transplant, LVRS, bullectomy, or lobectomy.
* Clinically significant bronchiectasis.
* Unable to safely discontinue anticoagulants or platelet activity inhibitors for 7 days.
* Uncontrolled pulmonary hypertension (systolic pulmonary arterial pressure >45mmHg) or evidence or history of CorPulmonale as determined by a recent echocardiogram (completed within the last 3 months prior to screening visit).
* Left ventricular ejection fraction (LVEF) less than 40% as determined by a recent echocardiogram (completed within the last 3 months prior to screening visit).
* Resting bradycardia (<50 bpm), Complex ventricular arrhythmia, sustained SVT.
* PaCO2 greater than 50mmHg on room air at screening.
* PaO2 less than 45mmHg on room air at screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-05-24 (Estimated)

PRIMARY OUTCOMES:
Prove that inter-lobar fissures can be completed to at least 95% in severe emphysema patients with previously failed bronchoscopic lung volume reduction | 2 years
  The investigators will determine that performing the surgery is feasible if the target inter-lobar fissure can be completed in at least 90% of the patients enrolled.
Incidence of severe adverse events | 2 years
  The investigators will actively monitor and record the severe adverse events that require any kind of additional intervention (medical or surgical) during and after the procedure. In case the treating physicians consider that the complications seen in patients outweigh the benefits obtained, the surgical technique will be revised and possible changes will be discussed.

SECONDARY OUTCOMES:
Percentage of patients to achieve target lung volume reduction | 2 years
  Describe the percentage of patients that achieve target lung volume reduction of at least 350mL at three months after the procedure.
Percentage of patients with quality of life improvement | 2 years
  Describe the changes in quality of life based on three subjective questionnaires that will be given to patients at baseline and three months after the intervention.
Percentage of patients with significant changes in pulmonary function testing | 2 years
  Describe the changes in PFTs after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheaton AG, Cunningham TJ, Ford ES, Croft JB; Centers for Disease Control and Prevention (CDC). Employment and activity limitations among adults with chronic obstructive pulmonary disease--United States, 2013. MMWR Morb Mortal Wkly Rep. 2015 Mar 27;64(11):289-95. PMID 25811677
- [Background] Global Initiative for Chronic Obstructive Lung Disease (GOLD): Global Strategy for the Diagnosis, Management, and Prevention of COPD 2022.
- [Background] Hartman JE, Vanfleteren LEGW, van Rikxoort EM, Klooster K, Slebos DJ. Endobronchial valves for severe emphysema. Eur Respir Rev. 2019 Apr 17;28(152):180121. doi: 10.1183/16000617.0121-2018. Print 2019 Jun 30. PMID 30996040
- [Background] Majid A, Kheir F, Alape D, Chee A, Parikh M, DeVore L, Agnew A, Gangadharan S. Combined Thoracoscopic Surgical Stapling and Endobronchial Valve Placement For Lung Volume Reduction With Incomplete Lobar Fissures: An Experimental Pilot Animal Study. J Bronchology Interv Pulmonol. 2020 Apr;27(2):128-134. doi: 10.1097/LBR.0000000000000617. PMID 31436607
- [Background] Celli BR, Wedzicha JA. Update on Clinical Aspects of Chronic Obstructive Pulmonary Disease. N Engl J Med. 2019 Sep 26;381(13):1257-1266. doi: 10.1056/NEJMra1900500. No abstract available. PMID 31553837
- [Background] Kochanek KD, Murphy S, Xu J, Arias E. Mortality in the United States, 2016. NCHS Data Brief. 2017 Dec;(293):1-8. PMID 29319473
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Background] Sullivan SD, Ramsey SD, Lee TA. The economic burden of COPD. Chest. 2000 Feb;117(2 Suppl):5S-9S. doi: 10.1378/chest.117.2_suppl.5s. PMID 10673466
- [Background] Rennard SI. COPD: overview of definitions, epidemiology, and factors influencing its development. Chest. 1998 Apr;113(4 Suppl):235S-241S. doi: 10.1378/chest.113.4_supplement.235s. PMID 9552012
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Maltais F. Exercise and COPD: therapeutic responses, disease-related outcomes, and activity-promotion strategies. Phys Sportsmed. 2013 Feb;41(1):66-80. doi: 10.3810/psm.2013.02.2001. PMID 23445862
- [Background] Fishman A, Martinez F, Naunheim K, Piantadosi S, Wise R, Ries A, Weinmann G, Wood DE; National Emphysema Treatment Trial Research Group. A randomized trial comparing lung-volume-reduction surgery with medical therapy for severe emphysema. N Engl J Med. 2003 May 22;348(21):2059-73. doi: 10.1056/NEJMoa030287. Epub 2003 May 20. PMID 12759479
- [Background] Fessler HE, Permutt S. Lung volume reduction surgery and airflow limitation. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):715-22. doi: 10.1164/ajrccm.157.3.9608004. PMID 9517581
- [Background] Naunheim KS, Wood DE, Krasna MJ, DeCamp MM Jr, Ginsburg ME, McKenna RJ Jr, Criner GJ, Hoffman EA, Sternberg AL, Deschamps C; National Emphysema Treatment Trial Research Group. Predictors of operative mortality and cardiopulmonary morbidity in the National Emphysema Treatment Trial. J Thorac Cardiovasc Surg. 2006 Jan;131(1):43-53. doi: 10.1016/j.jtcvs.2005.09.006. Epub 2005 Dec 5. PMID 16399293
- [Background] DeCamp MM Jr, McKenna RJ Jr, Deschamps CC, Krasna MJ. Lung volume reduction surgery: technique, operative mortality, and morbidity. Proc Am Thorac Soc. 2008 May 1;5(4):442-6. doi: 10.1513/pats.200803-023ET. PMID 18453353
- [Background] DeCamp MM, Blackstone EH, Naunheim KS, Krasna MJ, Wood DE, Meli YM, McKenna RJ Jr; NETT Research Group. Patient and surgical factors influencing air leak after lung volume reduction surgery: lessons learned from the National Emphysema Treatment Trial. Ann Thorac Surg. 2006 Jul;82(1):197-206; discussion 206-7. doi: 10.1016/j.athoracsur.2006.02.050. PMID 16798215
- [Background] Labarca G, Uribe JP, Pacheco C, Folch E, Kheir F, Majid A, Jantz MA, Mehta HJ, Patel N, Herth FJF, Fernandez-Bussy S. Bronchoscopic Lung Volume Reduction with Endobronchial Zephyr Valves for Severe Emphysema: A Systematic Review and Meta-Analysis. Respiration. 2019;98(3):268-278. doi: 10.1159/000499508. Epub 2019 May 22. PMID 31117102
- [Background] Sciurba FC, Ernst A, Herth FJ, Strange C, Criner GJ, Marquette CH, Kovitz KL, Chiacchierini RP, Goldin J, McLennan G; VENT Study Research Group. A randomized study of endobronchial valves for advanced emphysema. N Engl J Med. 2010 Sep 23;363(13):1233-44. doi: 10.1056/NEJMoa0900928. PMID 20860505
- [Background] Eberhardt R, Gompelmann D, Schuhmann M, Reinhardt H, Ernst A, Heussel CP, Herth FJF. Complete unilateral vs partial bilateral endoscopic lung volume reduction in patients with bilateral lung emphysema. Chest. 2012 Oct;142(4):900-908. doi: 10.1378/chest.11-2886. PMID 22459779
- [Background] Shah PL, Herth FJ. Current status of bronchoscopic lung volume reduction with endobronchial valves. Thorax. 2014 Mar;69(3):280-6. doi: 10.1136/thoraxjnl-2013-203743. Epub 2013 Sep 5. PMID 24008689
- [Background] Cetti EJ, Moore AJ, Geddes DM. Collateral ventilation. Thorax. 2006 May;61(5):371-3. doi: 10.1136/thx.2006.060509. PMID 16648350
- [Background] Koster TD, Slebos DJ. The fissure: interlobar collateral ventilation and implications for endoscopic therapy in emphysema. Int J Chron Obstruct Pulmon Dis. 2016 Apr 13;11:765-73. doi: 10.2147/COPD.S103807. eCollection 2016. PMID 27110109
- [Background] Koster TD, van Rikxoort EM, Huebner RH, Doellinger F, Klooster K, Charbonnier JP, Radhakrishnan S, Herth FJ, Slebos DJ. Predicting Lung Volume Reduction after Endobronchial Valve Therapy Is Maximized Using a Combination of Diagnostic Tools. Respiration. 2016;92(3):150-7. doi: 10.1159/000448849. Epub 2016 Aug 31. PMID 27577190
- [Background] Gompelmann D, Eberhardt R, Slebos DJ, Brown MS, Abtin F, Kim HJ, Holmes-Higgin D, Radhakrishnan S, Herth FJ, Goldin J. Diagnostic performance comparison of the Chartis System and high-resolution computerized tomography fissure analysis for planning endoscopic lung volume reduction. Respirology. 2014 May;19(4):524-30. doi: 10.1111/resp.12253. Epub 2014 Feb 25. PMID 24612306
- [Background] Herth FJ, Eberhardt R, Gompelmann D, Ficker JH, Wagner M, Ek L, Schmidt B, Slebos DJ. Radiological and clinical outcomes of using Chartis to plan endobronchial valve treatment. Eur Respir J. 2013 Feb;41(2):302-8. doi: 10.1183/09031936.00015312. Epub 2012 May 3. PMID 22556025
- [Background] Herth FJF, Slebos DJ, Criner GJ, Valipour A, Sciurba F, Shah PL. Endoscopic Lung Volume Reduction: An Expert Panel Recommendation - Update 2019. Respiration. 2019;97(6):548-557. doi: 10.1159/000496122. Epub 2019 Mar 5. PMID 30836374
- [Background] Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, Marciniuk DD, Denberg T, Schunemann H, Wedzicha W, MacDonald R, Shekelle P; American College of Physicians; American College of Chest Physicians; American Thoracic Society; European Respiratory Society. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91. doi: 10.7326/0003-4819-155-3-201108020-00008. PMID 21810710
- [Background] Slebos DJ, Shah PL, Herth FJ, Valipour A. Endobronchial Valves for Endoscopic Lung Volume Reduction: Best Practice Recommendations from Expert Panel on Endoscopic Lung Volume Reduction. Respiration. 2017;93(2):138-150. doi: 10.1159/000453588. Epub 2016 Dec 20. PMID 27992862